CLINICAL TRIAL: NCT04542902
Title: Non-coding RNAs Analysis of Eosinophil Subtypes in Asthma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Kestutis Malakauskas, Principal Investigator, Clinical Professor, Head of Laboratory, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: LAB-1/2020
Record Dates: First submitted 2020-08-25; First posted 2020-09-09 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-08

CONDITIONS: Allergic Asthma; Severe Eosinophilic Asthma
Keywords: Eosinophils subtypes; Non-coding RNA; Exosome
MeSH Terms: conditions — Pulmonary Eosinophilia | interventions — Antigens, Dermatophagoides; Blood Specimen Collection; Allergens

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Allergic asthma patients (Experimental): Allergic asthma patients and sensitization to house dust mites (D. pteronyssinus) allergen.
  Interventions: Biological: Dermatophagoides pteronyssinus allergen; Procedure: Blood sampling; Procedure: Bronchial challenge with allergen
- Severe eosinophilic asthma patients (Experimental)
  Interventions: Procedure: Blood sampling
- Healthy subjects as a control group (Active Comparator): Healthy subjects without allergic and other chronic respiratory diseases (control group).
  Interventions: Procedure: Blood sampling

INTERVENTIONS:
Biological: Dermatophagoides pteronyssinus allergen — Dermatophagoides pteronyssinus allergen is required to perform allergen bronchial challenge test.
  Arms: Allergic asthma patients
Procedure: Blood sampling — An amount of a person's blood taken from their body for use in medical.
Procedure: Bronchial challenge with allergen — Bronchial challenge is performed with D. pteronyssinus allergen. Measurements of differences in eosinophils activity after allergen challenge.
  Arms: Allergic asthma patients

SUMMARY:
Chronic airway inflammation rich in eosinophils is an important feature seen in asthma. Airway and blood eosinophilia is associated with increased rates of asthma exacerbations and more intense treatment.

Recently, the existence of two distinct eosinophils subtypes was revealed-lung-resident eosinophils (rEOS), which maturate independently to interleukin (IL) 5, with the primary function to maintain tissue homeostasis, and inflammatory eosinophils (iEOS), which mature in IL-5-dependent manner and are mainly involved in immune responses. Eosinophils' effect on the airway remodeling in asthma depends not only on the activity but also by their viable number in the lungs. Blood iEOS infiltrate the airways mainly after the environmental stimulus like allergen and leave the airways with bronchial secretions. However, rEOS reside lung tissue for their entire lifetime regulating local immunity. Blood rEOS and iEOS ratio alters in asthma, compared with healthy controls. It is known that the predominant eosinophils subtype in allergic asthma are iEOS, while rEOS are basic subtype in severe eosinophilic asthma patients, moreover, they are different in adhesive properties and survivability as well. Distinct biological properties allows to speculate about their different functions in asthma, however, there are still little information. Data about differently expressed microRNA (miRNA) profiles in eosinophils in asthma suggests, that eosinophils subtypes can be distinct in non-coding RNA (ncRNA) - microRNA (miRNA), piwi-interacting RNA (piRNA) and long non-coding RNA (IncRNA) profiles that could describe their role in asthma pathogenesis and act as biomarkers to discern asthma phenotypes.

DETAILED DESCRIPTION:
Asthma is not cured, and only well-balanced treatment can control the course and severity of the disease. Most clinical symptoms rise from aberrant chronic airway inflammation mostly eosinophilic. Eosinophils are terminally differentiated granulocytes that actively contribute to innate and adaptive inflammatory cascades through the production and release of diverse chemokines, cytokines, lipid mediators and other growth factors. IL-5 plays a fundamental role in eosinophils maturation in the bone marrow, their recruitment, and activation at sites of inflammation.

Historically eosinophils were described as a critical player in host defense, including parasites, viruses, fungi, or bacteria, giving them a destructive inflammatory cell label. However, it became clear that steady-state eosinophils can contribute to the immunoregulation and tissue homeostasis as well. Studies revealed that there are distinct eosinophils subtypes - immunoregulatory lung-resident eosinophils (rEOS) and inflammatory eosinophils (iEOS), involved in immune responses. Distinct eosinophils subtypes with different functions determines the separate treatment. There are still only a few studies describing distinct eosinophils subtypes in the lungs or blood. It is the beginning of a new promising research area for better individualized eosinophilic asthma treatment, moreover, other eosinophilic diseases as well.

Peripheral blood eosinophils studies are sufficiently relevant to the tissue eosinophils studies, as blood eosinophils are released into the bloodstream in a fully maturated form. Moreover, peripheral blood study could give additional information with possibilities to prevent eosinophils effects in the early stage, before migration to the airways. Furthermore, the existence of tissue-resident eosinophils in peripheral blood is confirmed and primary research for eosinophil subtypes surface markers was made according to the data of human blood eosinophils.

Data about differently differently expressed microRNA (miRNA) profiles in eosinophils in asthma suggests, that eosinophils subtypes can be distinct in non-coding RNA (ncRNA) - microRNA (miRNA), piwi-interacting RNA (piRNA) and long non-coding RNA (IncRNA) profiles that could describe their role in asthma pathogenesis and act as biomarkers to discern asthma phenotypes.

Researchers have plan to expand research by analyzing non-coding RNA (ncRNA) - miRNA, piRNA and lncRNA profiles of rEOS and iEOS as well as selected ncRNA signatures in blood plasma estimating their diagnostic value. Moreover, additional investigation of ncRNA in eosinophil-derived exosomes will provide important data about possible effect of eosinophils subtypes on airway remodeling via secreted ncRNA. ncRNAs are key regulators for gene transcription. However, there is evidence about their dysregulation in eosinophils during asthma. It will give important information about molecular signaling pathways that regulate the activity of distinct eosinophil subtypes during health and asthma, and provide the essential information about possible new therapeutic targets for their control. Additionally researchers will investigate the biological differences between rEOS and iEOS, including surface integrins and eosinophilopoietins receptors expression, adhesive properties, survivability, synthesized reactive oxygen species and apoptosis, as well as their effect on pulmonary structural cells physiological activity as proliferation, apoptosis, migration, contractility and proteins production, and will relate it with molecular signaling pathways, regulated by distinct expressed ncRNAs. ncRNAs can be stored in eosinophils exosomes and expressed to the surrounding environment. Information about ncRNAs in eosinophils-derived exosomes will demonstrate their function by affecting the other cells, especially after migration to airways. Moreover, ncRNAs are stable and resistant to blood RNases and differentially expressed in several pathologies. Researchers suppose that altered blood levels of ncRNAs could act as a possible new diagnostic biomarker in asthma.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 18-70 years;
* Allergic asthma and sensitization to house dust mites (D. pteronyssinus) allergen, approved with: 1) medical history and symptoms more than one year; 2) skin prick test positive for D. pteronyssinus (positive wheals are those exceeding 3 mm in diameter greater than the negative control); 3) positive bronchial challenge with methacholine or documented reversible bronchial obstruction;
* Severe eosinophilic asthma;
* Premenopausal women if pregnancy test is negative;
* Healthy subjects without allergic and other chronic respiratory diseases (control group);
* Participants who gave his/her informed written consent.

Exclusion Criteria:

* Asthma exacerbation 1 month prior to study;
* Clinically significant permanent allergy symptoms (ex. cat or dog dander induced allergy);
* Contraindications to perform an allergy skin test and/or bronchial provocation test: 1) active airway infection 1 month prior the study; 2) used medicaments: inhaled glucocorticoids intake 1 month prior the study, antihistamines intake 7 days prior the study; 3) short acting β2 agonists 12 hours prior the study; 4) long acting β2 agonists 2 days prior the study; 5) leukotriene receptor antagonists prior 14 days;
* Contraindications for epinephrine;
* Other significant mental and / or internal diseases and conditions, which could be as exclusion criteria due to the opinion of the researcher;
* Alcohol or narcotic abuse;
* Pregnancy;
* Breast-feeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Fold changes of ncRNA expression between eosinophils subtypes | From 6 to 12 months
  Validated ncRNA expression of rEOS and iEOS in severe and non-severe eosinophilic asthma patients and healthy subjects.
ncRNA levels in rEOS- and iEOS-derived exosomes | From 12 to 18 months
  Qualitative and quantitative selected ncRNA levels in rEOS- and iEOS-derived exosomes of all investigated groups.

SECONDARY OUTCOMES:
Fold changes of ncRNA profiles of distinct eosinophil subtypes | From 6 to 12 months
  Non-validated whole ncRNA profiles of distinct eosinophil subtypes in severe and non-severe eosinophilic asthma patients and healthy subjects.
The fold changes of rEOS and iEOS surface integrins expression | From 6 to 12 months
  The gene expression of selected outer-membrane integrins in eosinophil subtypes.
The fold changes of rEOS and iEOS eosinophilopoietins receptors expression | From 6 to 12 months
  The gene expression of interleukin (IL)-5, IL-3, and granulocyte-macrophage colony-stimulating factor in eosinophil subtypes.
The efficiency of iEOS and rEOS adhesion | From 6 to 12 months
  The differences in stable adhered iEOS and rEOS quantity in the combined cell culture with airway smooth muscle (ASM) cells or pulmonary fibroblasts compared between the investigated groups.
iEOS and rEOS survival differences | From 6 to 12 months
  Viable iEOS and rEOS number after an appropriate period of time in combined cell culture with ASM cells or pulmonary fibroblasts.
Quantity of iEOS and rEOS synthesized reactive oxygen species | From 6 to 12 months
  Relative differences between iEOS and rEOS synthesized reactive oxygen species quantity after an appropriate period of incubation alone or with ASM cells or pulmonary fibroblasts.
Apoptotic iEOS and rEOS number | From 6 to 12 months
  The number of apoptotic iEOS and rEOS after an appropriate period of time in combined cell culture with ASM cells or pulmonary fibroblasts.
Concentrations of iEOS and rEOS produced proteins in investigated subjects' body fluids. | From 6 to 12 months
  Selected iEOS and rEOS proteins concentrations, measured in investigated subjects body fluids, expressed as the amount of protein in the respective amount of fluid sample.
iEOS and rEOS effect on airway smooth muscle cells or pulmonary fibroblasts proliferation | From 6 to 12 months
  The quantity of ASM cells or pulmonary fibroblasts after several repeats of proliferation in the presence or absence of eosinophil subtypes.
iEOS and rEOS effect on apoptotic ASM cells and pulmonary fibroblasts number | From 6 to 12 months
  The number of apoptotic ASM cells and pulmonary fibroblasts after an appropriate period of time in combined cell culture with iEOS and rEOS.
iEOS and rEOS effect on migration of ASM cells. | From 6 to 12 months
  The migrated ASM cells number after an appropriate period of time in combined cell culture with iEOS and rEOS
iEOS and rEOS effect on migration of pulmonary fibroblasts | From 6 to 12 months
  The migrated pulmonary fibroblasts number after an appropriate period of time in combined cell culture with iEOS and rEOS
iEOS and rEOS effect on ASM cells contractility | From 6 to 12 months
  The relative efficiency of ASM cells' ability to contract collagen gel after an appropriate period of time in combined cell culture with iEOS and rEOS, expressed as reduced poured gel size in percentage, compared with control ASM cells without incubation with eosinophils.
iEOS and rEOS effect on pulmonary fibroblasts contractility | From 6 to 12 months
  The relative efficiency of pulmonary fibroblasts ability to contract collagen gel after an appropriate period of time in combined cell culture with iEOS and rEOS. expressed as reduced poured gel size in percentage, compared with control pulmonary fibroblasts, without incubation with eosinophils.
iEOS and rEOS effect on fold changes of ASM cells and pulmonary fibroblasts proteins expression; | From 6 to 12 months
  Altered selected ASM cells and pulmonary fibroblasts proteins expression, after incubation with iEOS and rEOS, expressed as fold changes in comparison with control cells, without incubation with eosinophils
iEOS and rEOS effect on fold changes of ASM cells and pulmonary fibroblasts proteins gene expression; | From 6 to 12 months
  Altered selected ASM cells and pulmonary fibroblasts proteins gene expression, after incubation with iEOS and rEOS, expressed as fold changes in comparison with control cells, without incubation with eosinophils

CONTACTS AND LOCATIONS:
Locations (1):
- Lithuanian University of Health Sciences, Pulmonology Department, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barnig C, Alsaleh G, Jung N, Dembele D, Paul N, Poirot A, Uring-Lambert B, Georgel P, de Blay F, Bahram S. Circulating Human Eosinophils Share a Similar Transcriptional Profile in Asthma and Other Hypereosinophilic Disorders. PLoS One. 2015 Nov 2;10(11):e0141740. doi: 10.1371/journal.pone.0141740. eCollection 2015. PMID 26524763
- [Background] Mazzeo C, Canas JA, Zafra MP, Rojas Marco A, Fernandez-Nieto M, Sanz V, Mittelbrunn M, Izquierdo M, Baixaulli F, Sastre J, Del Pozo V. Exosome secretion by eosinophils: A possible role in asthma pathogenesis. J Allergy Clin Immunol. 2015 Jun;135(6):1603-13. doi: 10.1016/j.jaci.2014.11.026. Epub 2015 Jan 21. PMID 25617225
- [Background] Mesnil C, Raulier S, Paulissen G, Xiao X, Birrell MA, Pirottin D, Janss T, Starkl P, Ramery E, Henket M, Schleich FN, Radermecker M, Thielemans K, Gillet L, Thiry M, Belvisi MG, Louis R, Desmet C, Marichal T, Bureau F. Lung-resident eosinophils represent a distinct regulatory eosinophil subset. J Clin Invest. 2016 Sep 1;126(9):3279-95. doi: 10.1172/JCI85664. Epub 2016 Aug 22. PMID 27548519
- [Background] Mitchell PS, Parkin RK, Kroh EM, Fritz BR, Wyman SK, Pogosova-Agadjanyan EL, Peterson A, Noteboom J, O'Briant KC, Allen A, Lin DW, Urban N, Drescher CW, Knudsen BS, Stirewalt DL, Gentleman R, Vessella RL, Nelson PS, Martin DB, Tewari M. Circulating microRNAs as stable blood-based markers for cancer detection. Proc Natl Acad Sci U S A. 2008 Jul 29;105(30):10513-8. doi: 10.1073/pnas.0804549105. Epub 2008 Jul 28. PMID 18663219
- [Background] Perry MM, Tsitsiou E, Austin PJ, Lindsay MA, Gibeon DS, Adcock IM, Chung KF. Role of non-coding RNAs in maintaining primary airway smooth muscle cells. Respir Res. 2014 May 16;15(1):58. doi: 10.1186/1465-9921-15-58. PMID 24886442
- [Background] Rodrigo-Munoz JM, Canas JA, Sastre B, Rego N, Greif G, Rial M, Minguez P, Mahillo-Fernandez I, Fernandez-Nieto M, Mora I, Barranco P, Quirce S, Sastre J, Del Pozo V. Asthma diagnosis using integrated analysis of eosinophil microRNAs. Allergy. 2019 Mar;74(3):507-517. doi: 10.1111/all.13570. Epub 2018 Oct 11. PMID 30040124
- [Background] Zhu Y, Mao D, Gao W, Han G, Hu H. Analysis of lncRNA Expression in Patients With Eosinophilic and Neutrophilic Asthma Focusing on LNC_000127. Front Genet. 2019 Mar 19;10:141. doi: 10.3389/fgene.2019.00141. eCollection 2019. PMID 30941157
- [Background] Weller PF, Spencer LA. Functions of tissue-resident eosinophils. Nat Rev Immunol. 2017 Dec;17(12):746-760. doi: 10.1038/nri.2017.95. Epub 2017 Sep 11. PMID 28891557
- [Background] Rosenberg HF, Dyer KD, Foster PS. Eosinophils: changing perspectives in health and disease. Nat Rev Immunol. 2013 Jan;13(1):9-22. doi: 10.1038/nri3341. Epub 2012 Nov 16. PMID 23154224
- [Background] Rothenberg ME, Hogan SP. The eosinophil. Annu Rev Immunol. 2006;24:147-74. doi: 10.1146/annurev.immunol.24.021605.090720. PMID 16551246